CLINICAL TRIAL: NCT02078375
Title: The PRESS RA Study: Protein and Resistance Exercise Supplementation Study for Rheumatoid Arthritis
Brief Title: The PRESS RA: Protein and Resistance Exercise Supplementation Study for Rheumatoid Arthritis
Acronym: PRESSRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); American College of Rheumatology Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NA_00088317; R03AG045081 (NIH)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Proteins; Whey Proteins; Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbohydrate supplement (Placebo Comparator): Participants will be enrolled in a twice weekly resistance exercise program. They will receive a carbohydrate supplement to take twice daily (once after exercise).
  Interventions: Dietary Supplement: Carbohydrate (Placebo); Other: Resistance Exercise Program
- Protein Supplementation (Experimental): Participants will be enrolled in a twice weekly resistance exercise program. They will receive a twice daily protein supplement (once after exercise).
  Interventions: Dietary Supplement: Protein; Other: Resistance Exercise Program

INTERVENTIONS:
Dietary Supplement: Protein — whey protein plus casein protein
  Other Names: whey protein plus casein protein
  Arms: Protein Supplementation
Dietary Supplement: Carbohydrate (Placebo) — The twice daily placebo will consist of a carbohydrate and a small amount of protein
  Arms: Carbohydrate supplement
Other: Resistance Exercise Program — All participants will be enrolled in an individually supervised twice weekly (for 16 weeks) resistance exercise program

SUMMARY:
This study will evaluate if the combination of resistance exercise and protein supplementation will increase muscle strength and muscle mass among older individuals with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This study proposes a randomized trial to evaluate a tailored 16-week resistance exercise program, in combination with protein supplementation, for older individuals with RA. The exercise protocol in this study is distinctive because it combines dynamic and isometric (static) resistance exercise performed on specialized equipment that can accommodate the range of motion limitations frequently encountered in the older RA population. This study will also begin to evaluate if additional benefit can be achieved with daily protein supplementation

ELIGIBILITY:
Inclusion Criteria:

* age 60-95 years
* diagnosis of rheumatoid arthritis
* willing to participate in twice weekly exercise sessions

Exclusion Criteria:

* cognitive impairment
* recent heart surgery (within past 12 months)
* severe kidney disease
* use of supplemental oxygen
* presence of pacemaker
* diabetes that requires insulin for management
* allergy to soy or milk

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Body composition | after 16 weeks
  measured by dual-energy X-ray absorptiometry (DEXA) (lean mass vs fat mass)
Muscle strength | after 16 weeks
  measured by hand grip and biodex

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L. Manno, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Campus, Baltimore, Maryland, United States